CLINICAL TRIAL: NCT05103722
Title: A Pilot Study of Combined Aerobic and Resistance Exercise Training in Metastatic Renal Cell Carcinoma
Brief Title: Combined Aerobic and Resistance Exercise Training in Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: J2174; IRB00292763 (Other: JHU IRB)
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Renal Cell Carcinoma Metastatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Experimental): Patients with metastatic renal cell carcinoma (RCC) who are receiving immune-checkpoint inhibitor therapy
  Interventions: Other: Combined Aerobic and Resistance Exercise Training

INTERVENTIONS:
Other: Combined Aerobic and Resistance Exercise Training — Participants receive personalized exercise plan for home-based two days of aerobic exercises (20-30-minutes) and two days of resistance exercises per week for 12 weeks. After completion of study intervention, participants will be assessed at the of study visit at Week 24.

SUMMARY:
The trial studies the effects of personalized home-based aerobic and resistance exercises on quality of life, changes in physical activity levels, and the change in inflammatory myokines with the exercise intervention in Interleukin 6 (IL-6), C-reactive Protein (CRP), Leptin, Transforming growth factor beta (TGF-beta), and Interferon (INF) gamma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of RCC
* Patients being treated with standard of Programmed cell death protein 1 (anti-PD-1) or anti-PD-L1 immune-checkpoint inhibitor-containing standard of care regimen including patients who are about to start treatment or have been on treatment for a maximum of 4 weeks prior to signing consent
* Metastatic Measurable disease, as defined by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 with a life expectancy ≥ six months
* Physically able to enroll in the exercise program as determined by the treating medical oncologist and after review by Physical medicine and rehabilitation physicians at Johns Hopkins
* Adequate bone marrow reserve and organ function measured within 28 days prior to administration of study treatment with the following key parameters:
* Hematological:

  * Absolute neutrophil count ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 109/L
  * Hemoglobin≥ 9.0 g/dL
* Renal:

  * Serum Creatinine ≤ 1.5 x the upper limit of normal (ULN) or Calculated Creatinine clearance ≥ 30mL/min
* Hepatic:

  * Total bilirubin ≤ 1.5 x ULN (Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled)
  * Serum Aspartate aminotransferase (AST) and serum Alanine aminotransferase (ALT) ≤ 2.5 x ULN (For patients with documented liver metastases AST and/or ALT ≤ 5 x ULN)

Exclusion Criteria:

* The presence of bone metastasis in the spine, pelvis, and lower limbs
* Currently physically active or moderately active as determined by Leisure Score Index of Godin Leisure-Time Exercise Questionnaire (GSLTPAQ)
* History of underlying cardiovascular, respiratory, musculoskeletal disease or joint problems that preclude moderate physical activity
* Known underlying uncontrolled brain metastatic lesions requires steroids therapy and/or radiotherapy
* Major surgery within four weeks prior to enrollment.
* Radiotherapy for RCC 28 days prior to week 1 day 1

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who adhere to the exercise intervention | 2 years

SECONDARY OUTCOMES:
Percentage of patients screened compared to patients enrolled | 2 years
Percentage of patients who remained in the study and didn't drop off the study after enrollment | 2 years
Change in HRQoL as measured by FACT-G Questionnaire | Baseline, Week 4, Week 8, Week 12 and Week 24
  There are 27 items in Functional Assessment of Cancer Therapy: General (FACT-G) questionnaire, and they are scored on a scale from 0 to 4; 0 being "Not at All", and 4 being "Very much".
The incidence of grade 3-5 toxicities as per CTCAE 5.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ged, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No